CLINICAL TRIAL: NCT06215430
Title: A Phase I, Open-label, Fixed-sequence, Drug Interaction Study to Investigate the Effect of Multiple Oral Doses of LOXO-305 on CYP1A2, CYP2C9, and CYP2C19 Substrates Using a Probe Drug Cocktail in Healthy Subjects
Brief Title: A Study of Effect of Multiple Doses of LOXO-305 on the Pharmacokinetics of Single Oral Doses of CYP1A2, CYP2C9, CYP2C19 Substrates in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20010; J2N-OX-JZNE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-15; First posted 2024-01-22 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine; Omeprazole; Warfarin; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Probe Drug Cocktail (Experimental): Participants received 200 milligrams (mg) caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet on Day 1.
  Interventions: Drug: Caffeine Tablet; Drug: Omeprazole capsule; Drug: Warfarin tablet
- Period 2: Pirtobrutinib + Probe Drug Cocktail (Experimental): Participants received oral dose of 200 mg Pirtobrutinib once daily (QD) from Day 6 to Day 19. On Day 15, Pirtobrutinib was co-administered with 200 mg caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet.
  There was a 5-day washout period between the probe drug cocktail on Day 1 (Period 1) and the first dose of Pirtobrutinib on Day 6 (Period 2).
  Interventions: Drug: Caffeine Tablet; Drug: Omeprazole capsule; Drug: Warfarin tablet; Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Caffeine Tablet — Administered orally.
Drug: Omeprazole capsule — Administered orally.
Drug: Warfarin tablet — Administered orally.
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727
  Arms: Period 2: Pirtobrutinib + Probe Drug Cocktail

SUMMARY:
The main purpose of this study is to evaluate the effect of LOXO-305 on single oral dose of caffeine cytochrome P450 1A2 (CYP1A2) substrate, S-warfarin (CYP2C9 substrate), and omeprazole (CYP2C19 substrate) when administered as multiple doses by collecting the blood samples and conducting the blood tests to measure how much LOXO-305 is in the bloodstream and how the body handles and eliminates LOXO-305 in adult healthy participants. The study will also evaluate the safety and tolerability of LOXO-305. The study will be conducted in two periods. Participants will stay in this study for up to 67 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m^2), inclusive.
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator.
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods.
* Must have comply with all study procedures, including the 23-night stay at the Clinical Research Unit (CRU) and follow-up phone call.

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor.
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (Days 1 - 5)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Started | 16 | 0
Received at Least 1 Dose of Study Drug | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Period 2 (Days 6 - 23)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Started | 0 | 16 (All 16 participants who completed the Period 1 received pirtobrutinib along with probe drug cocktail in Period 2.)
Received at Least 1 Dose of Study Drug | 0 | 16
Completed | 0 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug.
Groups:
- Overall Study Participants: * Period 1: Participants received 200 milligrams (mg) caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet on Day 1.
  * Period 2: Participants received oral dose of 200 mg Pirtobrutinib once daily (QD) from Day 6 to Day 19. On Day 15, Pirtobrutinib was co-administered with 200 mg caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet.
  * There was a 5-day washout period between the probe drug cocktail on Day 1 (Period 1) and the first dose of Pirtobrutinib on Day 6 (Period 2).
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to 24 Hours Post-Dose (AUC0-24): Caffeine
Description: Area under the concentration time curve (AUC) from hour 0 to 24 hours post-dose (AUC0-24) of caffeine was reported.
Time Frame: Period 1, Day 1 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose); Period 2, Day 15 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose)
Population: All participants who received a dose of study drug, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter could be computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Period 1: Probe Drug Cocktail: In period 1, Participants received 200 milligrams (mg) caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet on Day 1.
- Period 2: Pirtobrutinib + Probe Drug Cocktail: In Period 2, Participants received oral dose of 200 mg Pirtobrutinib once daily (QD) from Day 6 to Day 19. On Day 15, Pirtobrutinib was co-administered with 200 mg caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet.
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour*nanogram per milliliter (h*ng/mL) | 39100 (31.8) | 37400 (31.8)

2. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to 24 Hours Post-Dose (AUC0-24): Paraxanthine
Description: AUC0-24 of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: All participants who received a dose of study drug, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter could be computed. Here 'overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 4
h*ng/mL | 20600 (12.1) | 18600 (17.7)

3. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to 24 Hours Post-Dose (AUC0-24): Omeprazole
Description: AUC0-24 of Omeprazole was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 2000 (100.9) | 3120 (61.6)

4. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to 24 Hours Post-Dose (AUC0-24): Warfarin
Description: AUC(0-24) of Warfarin was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 7320 (19.7) | 7880 (18.3)

5. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to 24 Hours Post-Dose (AUC0-24): Pirtobrutinib
Description: AUC0-24 of Pirtobrutinib was reported.
Time Frame: Period 2, Day 15 (0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours Post dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16
h*ng/mL | 119000 (24.4)

6. Primary Outcome: Area Under the Concentration-time Curve (AUC), From Hour 0 to the Last Measurable Concentration (AUC0-t): Caffeine
Description: AUC from hour 0 to the last measurable concentration (AUC0-t) of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 39100 (31.8) | 37400 (31.7)

7. Primary Outcome: Area Under the Concentration-time Curve (AUC), From Hour 0 to the Last Measurable Concentration (AUC0-t): Paraxanthine
Description: AUC0-t of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 20600 (12.1) | 19400 (14.0)

8. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to the Last Measurable Concentration (AUC0-t): Omeprazole
Description: AUC0-t of Omeprazole was reported.
Time Frame: Period 1, Day 1 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours postdose); Period 2, Day 15 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 1990 (101.0) | 3110 (61.7)

9. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to the Last Measurable Concentration (AUC0-t): Warfarin
Description: AUC0-t of Warfarin was reported.
Time Frame: Period 1, Day 1 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours postdose); Period 2, Day 15 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 17300 (19.1) | 19200 (20.0)

10. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 to the Last Measurable Concentration (AUC0-t): Pirtobrutinib
Description: AUC0-t of Pirtobrutinib was reported.
Time Frame: Period 2, Day 15 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16
h*ng/mL | 119000 (24.4)

11. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 Extrapolated to Infinity (AUC0-inf): Caffeine
Description: AUC from hour 0 extrapolated to infinity (AUC0-inf) of Caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 42600 (39.7) | 40000 (37.5)

12. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 Extrapolated to Infinity (AUC0-inf): Paraxanthine
Description: AUC0-inf of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 4 | 4
h*ng/mL | 23100 (10.1) | 20300 (17.4)

13. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 Extrapolated to Infinity (AUC0-inf): Omeprazole
Description: AUC0-inf of omeprazole was reported.
Time Frame: as for outcome 8
Population: All participants who received a dose of study drug had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter could be computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 2000 (101.0) | 3120 (61.6)

14. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Hour 0 Extrapolated to Infinity (AUC0-inf): Warfarin
Description: AUC0-inf of Warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
h*ng/mL | 20100 (21.1) | 22400 (21.9)

15. Primary Outcome: Percentage Extrapolation for AUC0-inf (%AUCextrap): Caffeine
Description: AUC0-inf (%AUCextrap) of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
percentage of AUCextrap | 5.20 (130.6) | 4.17 (149.3)

16. Primary Outcome: Percentage Extrapolation for AUC0-inf (%AUCextrap): Paraxanthine
Description: AUC0-inf (%AUCextrap) of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 4 | 4
percentage of AUCextrap | 12.0 (58.3) | 7.45 (63.6)

17. Primary Outcome: Percentage Extrapolation for AUC0-inf (%AUCextrap): Omeprazole
Description: %AUCextrap of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
percentage of AUCextrap | 0.421 (84.3) | 0.302 (97.8)

18. Primary Outcome: Percentage Extrapolation for AUC0-inf (%AUCextrap): Warfarin
Description: %AUCextrap of Warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
percentage of AUCextrap | 13.1 (33.5) | 13.4 (32.7)

19. Primary Outcome: Apparent Systemic Clearance (CL/F): Caffeine
Description: CL/F for caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
Liter per hour (L/h) | 4.70 (39.7) | 5.00 (37.5)

20. Primary Outcome: Apparent Systemic Clearance (CL/F): Omeprazole
Description: CL/F of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
L/h | 20.0 (101.0) | 12.8 (61.6)

21. Primary Outcome: Apparent Systemic Clearance (CL/F): Warfarin
Description: CL/F of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
L/h | 0.497 (21.1) | 0.447 (21.9)

22. Primary Outcome: Apparent Systemic Clearance (CL/F): Pirtobrutinib
Description: CL/F of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Pirtobrutinib 200 mg QD + Probe Drug Cocktail: In Period 2, Participants received oral dose of 200 mg Pirtobrutinib once daily (QD) from Day 6 to Day 19. On Day 15, Pirtobrutinib was co-administered with 200 mg caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet.
Arm/Group | Pirtobrutinib 200 mg QD + Probe Drug Cocktail
Number analyzed (Participants) | 16
L/h | 1.68 (24.4)

23. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Caffeine
Description: Cmax of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
ng/mL | 5060 (17.6) | 4990 (14.5)

24. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Paraxanthine
Description: Cmax of Paraxanthine was reported.
Time Frame: Period 1, Day 1 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 postdose); Period 2, Day 15 (Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
ng/mL | 1200 (14.3) | 1150 (14.6)

25. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Omeprazole
Description: Cmax of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
ng/mL | 901 (58.0) | 1350 (42.3)

26. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Warfarin
Description: Cmax of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
ng/mL | 585 (26.1) | 595 (25.2)

27. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Pirtobrutinib
Description: Cmax of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16
ng/mL | 9430 (24.6)

28. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax): Caffeine
Description: Tmax of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 0.500 [0.500 to 1.00] | 0.750 [0.500 to 1.00]

29. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax): Paraxanthine
Description: Tmax of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 10.0 [6.00 to 24.0] | 8.01 [6.00 to 12.0]

30. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax): Omeprazole
Description: Tmax of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 2.00 [1.50 to 4.00] | 2.50 [1.50 to 4.00]

31. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax): Warfarin
Description: Tmax of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 1.50 [0.500 to 3.00] | 1.50 [0.250 to 3.00]

32. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax): Pirtobrutinib
Description: Tmax of Pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16
hour (h) | 2.50 [0.767 to 4.00]

33. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ): Caffeine
Description: λZ of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
1/hour (1/h) | 0.116 (37.8) | 0.127 (34.6)

34. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ): Paraxanthine
Description: λZ of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 4 | 4
1/hour (1/h) | 0.0966 (24.0) | 0.120 (21.8)

35. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ): Omeprazole
Description: λZ of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
1/hour (1/h) | 0.611 (48.4) | 0.578 (37.2)

36. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ): Warfarin
Description: λZ of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
1/hour (1/h) | 0.0160 (17.1) | 0.0165 (16.4)

37. Primary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F): Caffeine
Description: Vz/F of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
Litre (L) | 40.4 (16.8) | 39.4 (18.1)

38. Primary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F): Omeprazole
Description: Vz/F of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
Litre (L) | 32.8 (45.7) | 22.2 (33.6)

39. Primary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F): Warfarin
Description: Vz/F of Warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
Litre (L) | 31.0 (18.4) | 27.1 (21.0)

40. Primary Outcome: Metabolite to Parent Drug AUC Ratio (MRAUC): AUC Ratio of Paraxanthine to Caffeine
Description: AUC Ratio of paraxanthine (Metabolite) to caffeine (Parent drug) was reported.
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
Ratio | 0.528 (29.1) | 0.518 (27.8)

41. Primary Outcome: Mean Residence Time (MRT): Caffeine
Description: MRT of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 8.58 (35.8) | 8.03 (30.9)

42. Primary Outcome: Mean Residence Time (MRT): Paraxanthine
Description: MRT of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 4 | 4
hour (h) | 12.8 (18.3) | 10.9 (14.8)

43. Primary Outcome: Mean Residence Time (MRT): Omeprazole
Description: MRT of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 3.22 (32.4) | 3.58 (20.1)

44. Primary Outcome: Mean Residence Time (MRT): Warfarin
Description: MRT of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 56.8 (18.9) | 57.9 (18.7)

45. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2): Caffeine
Description: t1/2 of caffeine was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 5.96 (37.8) | 5.47 (34.6)

46. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2): Paraxanthine
Description: t1/2 of Paraxanthine was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 4 | 4
hour (h) | 7.17 (24.0) | 5.79 (21.8)

47. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2): Omeprazole
Description: t1/2 of omeprazole was reported.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 1.13 (48.4) | 1.20 (37.2)

48. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2): Warfarin
Description: t1/2 of warfarin was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Period 1: Probe Drug Cocktail | Period 2: Pirtobrutinib + Probe Drug Cocktail
Number analyzed (Participants) | 16 | 16
hour (h) | 43.2 (17.1) | 42.0 (16.4)

ADVERSE EVENTS:
Time Frame: From Baseline up to End of Study i.e. 30 days.
Description: All participants who had received at least 1 dose of study drug. Participants were classified into groups based on actual treatment received.
Groups:
- Probe Drug Cocktail: Participants received 200 milligrams (mg) caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet on Day 1.
- Pirtobrutinib 200 mg QD: Participants received oral dose of 200 mg Pirtobrutinib once daily (QD) from Day 6 to Day 19.
- Pirtobrutinib 200 mg QD + Probe Drug Cocktail: Participant received 200 mg Pirtobrutinib co-administered with 200 mg caffeine tablet, 40 mg omeprazole capsule, and 10 mg warfarin tablet as a single dose of probe drug cocktail, along with 10 mg vitamin K tablet on Day 15.
Arm/Group | Probe Drug Cocktail | Pirtobrutinib 200 mg QD | Pirtobrutinib 200 mg QD + Probe Drug Cocktail
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 8/16 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probe Drug Cocktail (N=16) | Pirtobrutinib 200 mg QD (N=16) | Pirtobrutinib 200 mg QD + Probe Drug Cocktail (N=16)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT06215430/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT06215430/SAP_001.pdf